CLINICAL TRIAL: NCT04213664
Title: Prognostic Value of Pretreatment Lymphocyte-to-monocyte Ratio in Patients With in Non-metastatic Renal Cell Carcinoma: a Systematic Review and Meta-analysis
Brief Title: Meta-analysis of the Prognostic Value of Lymphocyte to Monocyte Ratio (LMR) in Non-metastatic Renal Cell Carcinoma.
Acronym: LMR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Dario Garcia-Rojo, Principal Investigator, Corporacion Parc Tauli
Other Study IDs: CSPT-URO-2019; 2019/679 (Registry Identifier: Corporacion Parc Tauli)
Record Dates: First submitted 2019-12-25; First posted 2019-12-30 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Renal Cell Carcinoma; Progression; Lymphocyte Disorder; Monocytosis; Local Disease
Keywords: renal cancer; lymphocyte to monocyte ratio; non metastatic; prognosis; meta-analysis; nephrectomy
MeSH Terms: conditions — Carcinoma, Renal Cell; Disease Progression; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- non-metastatic renal cell carcinoma: Pretreatment lymphocyte to monocyte ratio in non-metastatic patients with renal cell
  Interventions: Other: prognosis

INTERVENTIONS:
Other: prognosis — cancer and overall survival cancer specific survival cancer and recurrence-free survival cancer and disease-free survival lymphocyte to monocyte ratio in non-metastatic renal cancer and progression-free survival

SUMMARY:
PubMed, ScienceDirect, Cochrane Database of Systematic Reviews will be used to search for articles published from January 1965 to July 2019 using the key words "renal cancer", "lymphocyte to monocyte ratio" and "prognosis". No restrictions to date, language, or article type will be applied. Cohort or observational studies in patients with non-metastatic renal cell carcinoma histopathologically confirmed, with hazard ratios (HR) and corresponding 95% confidence intervals (CI) that assessed association between LMR and overall survival (OS), cancer-specific survival (CSS), recurrence-free survival (RFS), and disease-free survival (DFS) will be analyzed.

DETAILED DESCRIPTION:
A systematic review of the literature will be carried out using Patient, Intervention, Comparison and Outcome method (PICO), with the aim of answering the following clinical question: "Is pretreatment under lymphocyte to monocyte ratio (LMR) a prognostic factor in non-metastatic renal cell carcinoma ? "

All analyzes will be based on previously published studies. For this reason, patient consent and ethical approval will not be required.

An exhaustive search will be conducted in PubMed, Science Direct and Cochrane Database of Systematic Reviews for eligible studies that explored the prognostic role of LMR in patients with localized renal tumors, who underwent to partial or radical nephrectomy from January 1965 to July 2019. The terms search will include: "monocyte lymphocyte ratio", "renal cancer", "prognosis".

Cohort studies or observational studies will be included, patients with localized renal tumors who underwent partial or radical nephrectomy, with histopathologically confirmed neoplasms, who had access to the full text and without language limitation.

Inclusion:

Any observational study (cross-sectional, case-control, longitudinal with cross-sectional data) will be included.

Patients with localized renal tumors who underwent partial or radical nephrectomy, with histopathologically confirmed neoplasms, who had access to the full text and without language limitation will be included.

Exclusion: Reviews, case reports, conference abstracts, letters, animal or cell studies.

Relevant articles will be identified in duplicate by two independent reviewers by first screening the titles and abstracts followed by the full text against inclusion and exclusion criteria. Any disagreement will be resolved by consensus with a third reviewer experienced in the renal cancer management.

The studies reflected the hazard ratio (HR) and corresponding 95% confidence intervals (CI), in which the overall survival (OS), specific cancer specific survival (CSS), recurrence-free survival (RFS), disease-free survival (DFS) and progression-free survival (PFP).

Information will be extracted for the first author, publication year, geographic location, study design, patient information (sample size, mean/median age, sex distribution, performance status), LMR, endpoint (OS, CSS, RFS, DFS, PFS), therapy, follow up duration, multivariate factors, hazard ratio (HR) and corresponding 95% confidence intervals (CIs), or exact P values. When univariate HR and multivariate HR were both reported, only the multivariate HR will be used.

OS is defined as the interval from the date of surgery in the primary tumor until death. CSS is defined as the interval from the date of surgery in the primary tumor to death for urological tumors. RFS is defined as the interval from the date of surgery in the primary tumor to local, regional or distant recurrence or death from any cause. DFS is defined as the interval from the date of surgery in the primary tumor to local, regional or distant recurrence. PFS is defined as the interval from the date of surgery in the primary tumor to the progression of the disease (including local recurrence or distant metastasis) or death.

The Newcastle-Ottawa Scale (NOS) will be used to assess the quality of studies. A maximum of 9 points can be given for each study in the categories of: selection of patients, comparability of the study groups, and assessment of outcomes. We will define high-quality studies with scores >7.

If the necessary data are available, subgroup analyses will be performed to explore the potential sources of heterogeneity according to country, analysis type, tumor type, sample size and cut-off value.

Statistical study:

Data will be combined using random effect models. The Cochrane χ² (Cochrane Q) statistic and the I² test will be used to analyze heterogeneity.

Before calculating the combined results for all trials, statistical heterogeneity will be evaluated by using the I² statistic and p-value, which assessed the appropriateness of pooling the individual study results. The I² value provided an estimate of the amount of variance across studies because of heterogeneity rather than chance. I² values of 25%, 50%, and 75% corresponded to low, moderate, and high levels of heterogeneity, respectively. If p> 0.05, the heterogeneity will be not substantial. Thus, a fixed-effect model will be used to calculate forest plots. If p < 0.05, however, the heterogeneity will be considered substantial. Then a random effects models were used.

The publication bias will be graphically explored through funnel plot, and Duval and Tweedie's "trim-and-fill" test will be used to correct possible publication bias.

Statistical significance was defined as p less than 0.05.

Statistics will done using R 3.5.0 (R Core Team, 2018) and the meta (v4.1-5; Schwarzer, Guido, 2019) package.

ELIGIBILITY:
Inclusion Criteria:

* PubMed, ScienceDirect, Cochrane Database of Systematic Reviews will be used to search for articles published from January 1965 to July 2019 using the key words "renal cancer", "lymphocyte to monocyte ratio" and "prognosis".
* No restrictions to date or language will be applied.
* Cohort or observational studies in patients with non-metastatic renal cell carcinoma who underwent radical or partial nephrectomy, with hazard ratios (HR) and corresponding 95% confidence intervals (CI) that assessed association between LMR and overall survival (OS), cancer-specific survival (CSS), recurrence-free survival (RFS), and disease-free survival (DFS) will be analyzed.

  * -There were no restrictions about gender and ethnicity.

Exclusion Criteria:

* Reviews, case reports, conference abstracts, letters, animal or cell studies.
* Patients were diagnosed non-metastatic renal cell carcinoma, but without standard treatments (Ablative therapy).
* Preoperative inflammatory markers were not measured.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-metastatic renal cell carcinoma who underwent radical or partial nephrectomy
Sampling Method: Non-Probability Sample
Enrollment: 4666 (Estimated)
Dates: Start 2019-12-31 (Actual); Primary Completion 2020-01-02 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Preoperative Lymphocyte to Monocyte Ratio ( LMR) is a prognostic factor in non-metastatic renal cell carcinoma | Preoperative Lymphocyte to Monocyte Ratio ( LMR) will be determined one month before surgical treatment. Follow-up: through study completion, an average of 5 years.
  Preoperative Lymphocyte to Monocyte Ratio ( LMR) is a prognostic factor patients who underwent nephrectomy for non-metastatic renal cell carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Garcia-Rojo, Principal Investigator — Corporacion Parc Tauli.Sabadell. Spain
Locations (1):
- Corporacion Parc Tauli, Sabadell, Outside U.S./Canada, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li J, Cheng Y, Ji Z. Prognostic value of pretreatment lymphocyte-to-monocyte ratio in patients with urologic tumors: A PRISMA-compliant meta-analysis. Medicine (Baltimore). 2019 Jan;98(2):e14091. doi: 10.1097/MD.0000000000014091. PMID 30633220
- [Background] Grimes N, Tyson M, Hannan C, Mulholland C. A Systematic Review of the Prognostic Role of Hematologic Scoring Systems in Patients With Renal Cell Carcinoma Undergoing Nephrectomy With Curative Intent. Clin Genitourin Cancer. 2016 Aug;14(4):271-6. doi: 10.1016/j.clgc.2016.01.006. Epub 2016 Jan 22. PMID 26949171
- [Background] Wang X, Su S, Guo Y. The clinical use of the platelet to lymphocyte ratio and lymphocyte to monocyte ratio as prognostic factors in renal cell carcinoma: a systematic review and meta-analysis. Oncotarget. 2017 Sep 20;8(48):84506-84514. doi: 10.18632/oncotarget.21108. eCollection 2017 Oct 13. PMID 29137443
- [Result] Hutterer GC, Stoeckigt C, Stojakovic T, Jesche J, Eberhard K, Pummer K, Zigeuner R, Pichler M. Low preoperative lymphocyte-monocyte ratio (LMR) represents a potentially poor prognostic factor in nonmetastatic clear cell renal cell carcinoma. Urol Oncol. 2014 Oct;32(7):1041-8. doi: 10.1016/j.urolonc.2014.04.001. Epub 2014 Jul 11. PMID 25027686
- [Result] Chang Y, Fu Q, Xu L, Zhou L, Liu Z, Yang Y, Lin Z, Xu J. Prognostic value of preoperative lymphocyte to monocyte ratio in patients with nonmetastatic clear cell renal cell carcinoma. Tumour Biol. 2016 Apr;37(4):4613-20. doi: 10.1007/s13277-015-4300-7. Epub 2015 Oct 27. PMID 26508025
- [Result] Xia WK, Wu X, Yu TH, Wu Y, Yao XJ, Hu H. Prognostic significance of lymphocyte-to-monocyte ratio and CRP in patients with nonmetastatic clear cell renal cell carcinoma: a retrospective multicenter analysis. Onco Targets Ther. 2016 May 9;9:2759-67. doi: 10.2147/OTT.S101458. eCollection 2016. PMID 27274272
- [Derived] Garcia-Rojo D, Prera A, Munoz-Rodriguez J, Oliva JC, Dominguez A, Prats J. Prognostic value of lymphocyte-to-monocyte ratio previously determined to surgery in patients with non-metastatic renal cell carcinoma: A systematic review and a prisma-compliant meta-analysis. Medicine (Baltimore). 2021 Jan 22;100(3):e24152. doi: 10.1097/MD.0000000000024152. PMID 33546029